CLINICAL TRIAL: NCT04896580
Title: The Benefits of Nature-based Walking for Breast Cancer Survivors: a Pilot Study
Brief Title: IIT2020-20-SHIRAZIP-WALK: Nature Walks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Celina Shirazipour, Assistant Professor, Cedars-Sinai Cancer Research Center for Health Equity, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00001356
Record Dates: First submitted 2021-04-19; First posted 2021-05-21 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Cancer; Lymphoma; Leukemia; Prostate Cancer; Thyroid Cancer; Hematologic Malignancy; Non-hodgkin Lymphoma
Keywords: Nature; Exercise; Walking; Psychosocial Well-Being
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Lymphoma; Leukemia; Prostatic Neoplasms; Thyroid Neoplasms; Hematologic Neoplasms; Lymphoma, Non-Hodgkin; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active (Experimental): Participants will be asked to complete a 12 week exercise program
  Interventions: Behavioral: Nature based exercise

INTERVENTIONS:
Behavioral: Nature based exercise — Participants will engage in three months of moderate intensity PA, consisting of three 50-minute walking sessions per week (5-minute warm-up, 40 minute walk, 5 minute cool-down and stretch) with an exercise physiologist for 12 weeks.

SUMMARY:
The purpose of this study is to examine whether nature-based activities provide benefits for breast cancer survivors. The investigators want to know whether a nature-based exercise program is feasible. Women who were diagnosed with breast cancer and have completed cancer treatment will be recruited for the main study. The main study will enroll up to 20 breast cancer subjects in total.

This intervention will also include a sub-study examining the same outcomes among adolescents and young adult (AYA) subjects who were diagnosed with cancer (any type) and have completed cancer treatment. The sub-study will enroll up to 20 AYA (ages 18-39) subjects.

DETAILED DESCRIPTION:
This is a single-arm pilot study

MAIN STUDY Breast cancer survivors (n=20) will engage in three months of moderate intensity walking sessions three times a week in a nature and park conservation area. All walks will be supervised by certified clinical Exercise Physiologists (EP). Participants will be encouraged to keep the same days and walk session times throughout the intervention.

Sessions will be 50-minutes in total (5-minute warm-up, 40 minute walk, 5 minute cool-down and stretch). Session intensity will be tracked with Fitbits. Participants will be asked to reach a moderate intensity heart rate, defined as 40%-59% heart rate reserve.

Participants will complete surveys, physical assessments and collection of biomarkers at baseline and at end of study. Participants also have the option to participate in a 1 hr qualitative exit interview about their participation experiences.

Note. Based on any COVID pandemic restrictions at the time of a walk, sessions will be socially distanced one-on-one with an EP. When no restrictions are in place, they will take place in small groups (3-5 participants).

SUB-STUDY Adolescent and young adult (AYA) (ages 18-39) survivors (n=20) will complete all of the components of the Main-Study described above.

ELIGIBILITY:
Main Breast Cancer Study Inclusion Criteria:

1. Female previously diagnosed with breast cancer (clinical stages 1 - 3)
2. Minimum of 3 months post-active treatment completion
3. Maximum of 21 months post-active treatment completion
4. Physically able to complete baseline fitness assessments (e.g., 6-minute walk test, hand grip test, 1 RM leg press)
5. Ambulatory without assistance

Main Breast Cancer Study Exclusion Criteria:

1. Active treatment planned within the next 6 months.
2. Known metastatic disease.
3. Currently meeting physical activity guidelines (score of >23 on Godin-Shephard Leisure-Time Physical Activity Questionnaire).
4. Known allergy to Fitbit device or otherwise unable to wear Fitbit device.

Sub-study AYA Inclusion Criteria:

1. Men and women between age of 18 to 39
2. Previously diagnosed with cancer
3. Same inclusion criteria as the main study

Sub-Study AYA Exclusion Criteria:

1. Below 18 years old
2. Above 39 years old
3. Same Exclusion criteria as the main study except for no activity level cutoff score on Godin-Shephard Leisure-Time Physical Activity Questionnaire

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Number of participants that adhere to a 3-month nature-based walking program | 12 weeks
  Feasibility of Nature Walk Programs

SECONDARY OUTCOMES:
Short-term effects of green space and nature physical activity environments on well-being | Measured at Baseline and at Week 12
  PROMIS-29
Short-term effects of green space and nature physical activity environments on social well-being | Measured at Baseline and at Week 12
  PROMIS Social Support
Short-term effects of green space and nature physical activity environments on post-trauma growth and self-improvement | Measured at Baseline and at Week 12
  PTGI
Short-term effects of green space and nature physical activity environments on physical, social/family, emotional, and functional well-being | Measured at Baseline and at Week 12
  FACT-G
Biologic aging markers | Measured at Baseline and at Week 12
  DNA methylation, aging genes
TNF-α cytokine | Measured at Baseline and at Week 12
  TNF-α
Inflammatory cytokines | Measured at Baseline and at Week 12
  IL-1ß
Inflammatory cytokines, anti-inflammatory myokines | Measured at Baseline and at Week 12
  IL-6
Inflammatory marker | Measured at Baseline and at Week 12
  CRP
TGF-ß cytokine | Measured at Baseline and at Week 12
  TGF-ß
Anti-inflammatory cytokine | Measured at Baseline and at Week 12
  IL-10
IL-13 cytokine | Measured at Baseline and at Week 12
  IL-13

CONTACTS AND LOCATIONS:
Overall Officials: Celina Shirazipour, PhD, Principal Investigator — Cedars-Sinai Medical Center; Arash Asher, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shirazipour CH, Raines C, Liu E, Ruggieri RM, Capaldi JM, Luna-Lupercio B, Diniz MA, Gresham G, Bhowmick N, Haile RW, Asher A. Benefits of nature-based walking for breast cancer survivors. BMJ Open. 2023 Jun 16;13(6):e071041. doi: 10.1136/bmjopen-2022-071041. PMID 37328178